CLINICAL TRIAL: NCT01522027
Title: Use of Nerve Stimulation Technology to Aid in Percutaneous Tracheostomy in Intensive Care Patients.
Brief Title: Electrically Guided Needle Insertion: ICU Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro000026880
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2014-12

CONDITIONS: Percutaneous Tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nerve stimulator (Experimental): Twenty ICU patients will receive percutaneous tracheostomy via insertion of a needle/catheter connected to a nerve stimulator.
  Interventions: Procedure: Percutaneous tracheostomy

INTERVENTIONS:
Procedure: Percutaneous tracheostomy — Twenty ICU patients will receive percutaneous tracheostomy via insertion of a needle/catheter connected to a nerve stimulator.

SUMMARY:
Critically ill patients or patients under prolonged unconsciousness need a tube inserted into their windpipe to provide oxygen. This tube, called a tracheostomy tube, can be connected to a ventilation device to allow the patient to breathe when they cannot do it for themselves. In the hospital, doctors will perform a percutaneous tracheostomy (PT), where a needle is inserted through the skin of the neck into the windpipe, providing a guide for a tube that will dilate the tissue and create a hole that the tracheostomy tube can be inserted into. Although this is a common procedure in critical care units, it does carry some risks to the patient and is not always successful. The needle may puncture the back or side of the windpipe if it is inserted too far, or it can miss the windpipe altogether, causing damage to surrounding structures. We believe that doctors who perform PT would benefit from a method that improves the success rate of the procedure. We wish to test a device that alerts the doctor performing PT to when the needle tip is in the air-filled windpipe. The device has been proven to aid needle insertion in cadavers, but it needs to be tested on live patients. Since many intensive care patients undergo PT, we wish to test our technique on this population. It will be a controlled environment and the clinicians are experienced in PT. This technique should save valuable time, result in more accurate needle insertion, and lessen the risk of damaging other structures and tissues in the neck.

DETAILED DESCRIPTION:
Background: Critically ill patients occasionally require a tracheostomy tube to breathe. A percutaneous tracheostomy can be performed, where a needle/catheter is inserted into the trachea, followed by insertion of a guidewire and a tube that dilates the tissue, creating a hole for the tracheostomy tube. Although this is a common procedure, it does pose risks to the patient, including accidental puncture of nearby structures. We wish to test a device that alerts the doctor to when the needle tip is in the tracheal lumen. The device has been proven to aid needle insertion in cadavers, but it needs to be tested on live patients. Since many intensive care patients undergo PT, we wish to test our technique on this population.

Study objective: To evaluate the effectiveness of a nerve stimulator in aiding needle tracheostomy in live patients.

Hypothesis: Nerve stimulation equipment will help the physician guide and insert the needle tip into the tracheal lumen faster and with more accuracy than conventional techniques.

Primary outcome: speed and accuracy of needle tip placement in the trachea.

Procedure: This study will involve recruiting consenting adult patients from the University of Alberta Hospital General Systems Intensive Care Unit (ICU) who require percutaneous tracheostomy to insert a tracheal tube. In this population, a tracheostomy is usually performed as a means to provide long-term assisted ventilation without the need for endotracheal intubation. Briefly, the patient is sedated, the skin on their neck disinfected, and a local anesthetic injected into the anterior neck. A bronchoscope is inserted down the endotracheal tube to aid in visualization and localization of needle puncture. The cricothyroid membrane is located by palpating the anterior neck and an incision is made over the membrane. A small needle is inserted through the membrane to act as a guide for a larger needle-catheter assembly. Both needles are removed and a guidewire is inserted through the catheter. Using forceps, the insertion site is widened and a tube to dilate the opening is inserted. The tracheostomy tube is then inserted and the dilation tube and guidewire are removed. The endotracheal tube is removed and the ventilation apparatus is connected to the tracheostomy tube.

We will supply ICU physicians with a commonly used nerve stimulator (Stimuplex HNS 12, B.Braun, Germany) to attach to the needle-catheter assembly used to make the first insertion into the trachea. The nerve stimulator will be connected to a current meter, and a ground electrode will be attached to the body. When the needle tip is in contact with body tissue (i.e., tracheal wall), the electrical circuit will be closed, producing a reading of 1.0 mA on the current reader. Suspension of the needle tip in the airway will interrupt the circuit, producing a reading of 0.0 mA. In addition, an audible signal built into the nerve stimulator will alert the user to a change in current, warning that the needle tip has advanced too far and is in contact with the posterior or lateral tracheal wall.

The physician will perform percutaneous tracheostomy on 20 ICU patients that require endotracheal extubation and insertion of a tracheostomy tube. This will help support our preliminary observations which showed that the nerve stimulator was helpful in guiding needle insertion using human cadavers. By showing that the technique is equally as effective when used on live patients, we can argue that a nerve stimulator or similar device can ensure accurate, quick, and safe needle insertion when accessing the airway percutaneously.

Inclusion criteria: Adult; requires tracheostomy

Exclusion criteria: Failure to provide consent; known upper airway pathologies; known oro-pharyngeal or laryngeal disease, including any swelling, tumour, or infection; previous radiotherapy or operations on the neck; cervical spine fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 yrs)
* Requires tracheostomy

Exclusion Criteria:

* Failure to provide consent
* Known upper airway pathologies
* Known oro-pharyngeal or laryngeal disease, including any swelling, tumour, or infection
* Previous radiotherapy or operations on the neck
* Cervical spine fractures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Speed and accuracy of needle tip placement in the tracheal lumen | From positioning of the patient to withdrawal of needle; approximately 5 minutes
  The speed and accuracy with which a needle/catheter assembly connected to a nerve stimulator is inserted through the cricothyroid membrane into the tracheal lumen will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Tsui, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada